CLINICAL TRIAL: NCT03272048
Title: Identifying Effective Approaches to Counseling on Firearm Safety: A Randomized Experimental Design Among Firearm-familiar Individuals at Risk for Suicide
Brief Title: Identifying Effective Approaches to Counseling on Firearm Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Ian Stanley, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017.20703
Record Dates: First submitted 2017-08-30; First posted 2017-09-05 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Suicide
Keywords: Firearms
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low-Fear/Not-Temporary (Experimental)
  Interventions: Behavioral: Lethal Means Counseling
- Low-Fear/Temporary (Experimental)
  Interventions: Behavioral: Lethal Means Counseling
- High-Fear/Not-Temporary (Experimental)
  Interventions: Behavioral: Lethal Means Counseling
- High-Fear/Temporary (Experimental)
  Interventions: Behavioral: Lethal Means Counseling

INTERVENTIONS:
Behavioral: Lethal Means Counseling — Lethal means counseling is broadly defined as clinician-initiated discussions that encourage an individual at risk for suicide to safely store his or her firearms. Examples in this domain include applying a gun lock, separating the gun from its ammunition, dismantling the firearm and keeping its components locked and/or separated, or safely transferring the firearm to a trusted loved one, friend, or police station until risk abates (Bryan, Stone, & Rudd, 2011; Jin, Khazem, & Anestis, 2016). Further, given that recent purchasers of firearms are at markedly increased risk of death by suicide (Wintemute, Parham, Beaumont, Wright, & Drake, 1999), anticipatory counseling on firearm safety should also be considered for at-risk individuals who do not report currently owning or having access to a firearm, but who report prior firearm ownership/access or intentions of obtaining a firearm in the future (Harvard T.H. Chan School of Public Health, 2017).

SUMMARY:
Each year in the United States (U.S.), over 40,000 individuals die by suicide, and approximately half of these deaths occur by intentional, self-inflicted gunshot wounds. Given these staggering statistics, efforts to minimize individuals' access to firearms during at-risk periods has been identified as a critical if fraught suicide prevention strategy. Among individuals at risk for suicide who present to clinical settings, a crucial component of the clinical management of suicide risk is to ask about firearm ownership/access and counsel on firearm safety (e.g., encourage an at-risk person to transfer the firearm to a loved one until risk abates). Despite the clinical, ethical, and in some cases legal mandate of this intervention, a substantial proportion of clinicians are woefully undertrained and therefore unprepared to manage suicide risk and appropriately deliver counseling on firearm safety. Clinical and empirical evidence suggests that even among patients identified to be at increased risk for suicide, few clinicians ask about firearms or provide counseling on firearm safety. One key reason for this fissure between recommendations and actual implementation of recommendations is that strategies for discussing firearm safety in a way that is impactful and yields patient adherence to recommendations have yet to be established.

One common approach to attempt to garner pro-health behavior change is the use of fear appeals; however, research on the utility of this approach across non-firearm-related health interventions has been equivocal. Given the cultural importance placed on firearms in the U.S., the investigators contend that fear-based approaches to lethal means counseling may be counter-productive by creating defensive avoidance, thereby detracting from the purpose of counseling on firearm safety (i.e., patient safety).

Further, patient adherence to recommendations to limit access to a firearm during at-risk periods may be increased when clinicians emphasize that limits on firearm access will decline when suicide risk abates (i.e., limits on firearm access will likely not be permanent). However, research has yet to determine if varying the level of fear messaging and/or emphasis on temporariness is actually useful and acceptable.

To address this gap, the investigators will randomly assign participants to one of four experimental conditions: (1) low-fear/not-temporary; (2) low-fear/temporary; (3) high-fear/not-temporary; and (4) high-fear/temporary. Participants include undergraduate students who are vulnerable to suicide and reported owning or previously owning a firearm, reported access to a firearm, or reported possibly obtaining a firearm in the future. The investigators hypothesized that individuals randomly assigned to the low-fear/temporary group will (1) report greater intentions to adhere to recommendations to limit access to firearms during at-risk periods than the other groups at both post-intervention and one-month follow-up; (2) report greater actual adherence to recommendations at one-month follow-up; and (3) rate the lethal means counseling session as more acceptable than the other groups. Exploratory aims examined if the effects differed for individuals reporting actual current firearm ownership or access, membership in the National Rifle Association (NRA) or a similar organization, political affiliation, political ideology, greater personal importance of the Second Amendment, or severity of suicidal symptoms. Findings have the potential to inform clinical and public health approaches to limit at-risk individuals' access to firearms for safety purposes.

ELIGIBILITY:
Inclusion Criteria:

* Lifetime history of suicidal ideation or a suicide attempt
* Firearm familiarity (based on participants' self-report that they currently own a firearm, previously owned a firearm, have access to a firearm, have a desire to obtain a firearm in the future, or intend to obtain a firearm in the future)

Exclusion Criteria:

* Younger than 18 years old
* Imminent risk of harm to self or others necessitating hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Self-Reported Intentions to Adhere to Clinician Recommendations Scale | Change from Pre-Intervention to (a) Immediately Post-Intervention (i.e., assessed within minutes of completing the intervention) and (b) One-Month Follow-Up
Actual Adherence to Clinician Recommendations Scale | Change from Pre-Intervention to One-Month Follow-Up
Client Satisfaction Questionnaire | Immediately Post-Intervention (i.e., assessed within minutes of completing the intervention)
Credibility and Expectancy Questionnaire | Immediately Post-Intervention (i.e., assessed within minutes of completing the intervention)
Readiness to Change Scale | Change from Pre-Intervention to (a) Immediately Post-Intervention (i.e., assessed within minutes of completing the intervention) and (b) One-Month Follow-Up

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University Department of Psychology, Tallahassee, Florida, United States

REFERENCES:
- [Derived] Stanley IH, Hom MA, Sachs-Ericsson NJ, Gallyer AJ, Joiner TE. A pilot randomized clinical trial of a lethal means safety intervention for young adults with firearm familiarity at risk for suicide. J Consult Clin Psychol. 2020 Apr;88(4):372-383. doi: 10.1037/ccp0000481. Epub 2020 Jan 9. PMID 31916797